CLINICAL TRIAL: NCT03407755
Title: Air Versus SF6 for Descemet's Membrane Endothelial Keratoplasty (DMEK)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Mark Alberti, Principal Investigator, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-17006354
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Fuchs' Endothelial Dystrophy; Bullous Keratopathy
Keywords: Intraocular gas; Positioning; DMEK; Endothelial keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy

STUDY DESIGN:
Intervention Model Description: Patients randomized to either air or sulfur hexafluoride (SF6)
Who Masked: Participant, Investigator
Masking Description: Surgeon and patient masked to choice of intraocular gas. Study coordinator not masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Air (Active Comparator): Intraocular 100% atmospheric air (anterior chamber).
  Interventions: Procedure: Intraocular gas
- SF6 (Experimental): Intraocular 20% sulphur hexaflouride (anterior chamber).
  Interventions: Procedure: Intraocular gas

INTERVENTIONS:
Procedure: Intraocular gas — Participants randomized to either air or SF6 gas in the anterior chamber.

SUMMARY:
This blinded, randomized study compares the use of air and sulfur hexaflouride (SF6) tamponade in Descemet Membrane Endothelial Keratoplasty.

ELIGIBILITY:
Inclusion Criteria:

- Eligible for DMEK surgey

Exclusion Criteria:

Related to ocular health

* Re-DMEK or prior penetrating keratoplasty
* Ocular hypertension resistant to topical medication
* Previous vitrectomy
* Minimally invasive glaucoma devices
* Aphakia
* Anterior chamber or iris claw lens
* Implantable Collamer Lens (ICL)
* Clinically significant corneal scarring
* Central corneal thickness >750 µm
* BCVA < 0.1

Related to general health

* Not able to give informed consent
* Inability to position correctly due to organic or psychological condition.

Related to surgical procedure

* Graft diameter >9 mm or < 7mm
* Graft central endothelial cell count < 2000 cells/mm2
* Graft unfolding duration >1 hour
* Graft morphology grade 4-5
* Significant graft decentration (graft contour not visible in microscope)
* Significant presence of Descemet remnants in the graft-host interface
* Presence of inward folds
* Graft 'stroma-surface' placed facing away from recipient stroma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-05-01 (Estimated)

PRIMARY OUTCOMES:
Graft detachment | Occurence within 3 months postoperative
  Significant graft detachment: 1/3 of graft and affecting visual function. Measured by OCT.

SECONDARY OUTCOMES:
Visual acuity | 3 months postoperative
  Snellen chart (logMAR)
Gas fill | Serial measurements during postoperative week 1.
  Postoperative gas fill measured by OCT.
Positioning | 72 hours postoperative
  Pitch and roll of head using positioning device
Complications | Occurence within 3 months postoperative
  Any adverse outcome affecting the eye

CONTACTS AND LOCATIONS:
Overall Officials: Mark Alberti, MD, Study Director — Glostrup University Hospital, Copenhagen
Locations (1):
- Glostrup Hospital, University of Copenhagen, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
If permitted by the Danish Data Protection Agency